CLINICAL TRIAL: NCT04795960
Title: Microbiome Modification to Enhance Stelara Response in Crohn's Disease
Acronym: MIM-TESRIC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of eligible and interested patients
Sponsor: University of Michigan (Other)
Collaborators: Kenneth Rainin Foundation (Unknown)
Responsible Party: Principal Investigator, Peter Higgins, Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00185677
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Crohn Disease
Keywords: Ustekinumab; Stelara; Diet; Crohn's
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low serine diet (Experimental)
  Interventions: Dietary Supplement: Low serine diet
- High serine diet (Experimental)
  Interventions: Dietary Supplement: High serine diet

INTERVENTIONS:
Dietary Supplement: Low serine diet — Participants will be on this diet 1 week prior to initiation and 1 week after initiation of Ustekinumab (standard of care medication). The meals will be prepared in the Michigan Clinical Research Unit (MCRU) at the University of Michigan Health System and given to the participants.
  Arms: Low serine diet
Dietary Supplement: High serine diet — Participants will be on this diet 1 week prior to initiation and 1 week after initiation of Ustekinumab (standard of care medication). The meals will be prepared in the Michigan Clinical Research Unit (MCRU) at the University of Michigan Health System and given to the participants.
  Arms: High serine diet

SUMMARY:
This pilot study is being completed to determine whether a low-serine diet vs a high serine diet will reduce inflammation and symptoms in Crohn's disease (CD), as well as determine whether a low-serine diet (vs. a high serine diet) will improve responses in patients initiating therapy with Ustekinumab (Stelara), an FDA-approved biologic therapy for Crohn's disease.

DETAILED DESCRIPTION:
Eligible participants that will be given Ustekinumab as part of their standard of care will be enrolled in this study.

The study hypotheses include that a low serine diet (compared to a high serine diet) in patients with active CD will:

* Reduce the relative abundance of Adherent invasive ecoli (AIEC), and increase the relative abundance of Bacteroides and Faecalibacterium in stool of patients with Crohn's disease.
* Make patients more likely to respond to ustekinumab (anti-Interleukin12/23) therapy with control of inflammation as measured by the mean Simple endoscopic subscore Crohn's disease (SES-CD) in each group at week 25.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Crohn's Disease (CD) for at least 3 months prior to baseline. Appropriate documentation of biopsy results consistent with the diagnosis of CD, as determined by the investigator.
* Simple endoscopic subscore Crohn's disease (SES-CD) ≥ 7 for ileocolonic CD (or >=4 if only ileal CD) as confirmed by Dr. Higgins' scoring of colonoscopy.
* Are scheduled to begin Ustekinumab within the next 7-60 days
* Must be scheduled for clinically indicated colonoscopy, ordered by primary Gastroenterologist physician, and covered by insurance
* Must have access to a computer capable of completing video visits
* Must be willing to follow assigned meat-free diet provided by the study exclusively for 2 weeks
* Patients on anti-diarrheals must be on a stable dose for at least 2 weeks
* Prednisone is allowed up to a daily dose of 20 mg, with a stable dose for at least 1 week

Exclusion Criteria:

* Subject with a current diagnosis of Ulcerative Colitis
* Subjects requiring or receiving any Total Parenteral Nutrition (TPN) and/or exclusive enteral nutrition.
* Subjects who are pregnant or plan to become pregnant over the duration of the study
* Antibiotics in the previous 2 weeks.
* Probiotics in the previous 2 weeks.
* Ongoing therapy with infliximab, adalimumab, certolizumab, vedolizumab, or tofacitinib, is not allowed - must stop at least 1 week prior to ustekinumab start.
* Changes in dose of 5-aminosalicylates within the past 1 week - must be on a stable dose for at least one week.
* Changes in dose of immunomodulators (including Azathioprine, 6-mercaptopurine, methotrexate) within the past 4 weeks - must be on a stable dose for 4 weeks.
* Subjects with the following known complications of CD; Toxic megacolon, Short bowel syndrome or short gut (less than 100 centimeters, Ostomy, Symptomatic bowel strictures (scope cannot be passed through), any diagnosis that could interfere with nutrient absorption, note that actively draining fistulas are allowed at entry.
* Diabetes
* Subjects who use dietary supplements such as liquid or powder protein drinks/shakes, meal replacement shakes, and fiber supplements, etc. must be willing to stop at least 24 hours prior to starting the assigned diet
* Known allergy to soy products
* Oral Iron must be stopped at least 24 hours prior to baseline
* For severe anemia, intravenous (IV) iron can replace oral iron if approved and ordered by the prescribing physician
* Any subject currently hospitalized
* Any subject with a positive Clostridium difficile test (within 30 days of baseline) or currently being treated for Clostridium difficile.
* History of clinically significant medical condition or any other reason which, in the opinion of the PI, would interfere with the subject's participation
* Any active, chronic or recurrent infection that, based on the investigator's clinical assessment, makes the subject an unsuitable candidate for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-18 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
The mean simple endoscopic subscore Crohn's disease (SES-CD) score at week 25 between the two treatment groups. | 25 weeks
  This will be calculated by endoscopist at week 25.

SECONDARY OUTCOMES:
The mean Crohn's disease patient report outcomes (CD-PRO) score at week 2 will be compared between the two groups with Student's t test | 2 weeks
  There are a series of 52 questions to measure the extent of participant's crohn's disease. The higher the score the worse the disease.
The mean CD-PRO scores calculated by study team at week 25 will be compared between the two groups with Student's t test. | 25 weeks
  There are a series of 52 questions to measure the extent of participant's crohn's disease. The higher the score the worse the disease.

OTHER OUTCOMES:
The mean stool flagellin content at week 2 will be compared between the two groups with Student's t test. | 2 weeks
  This will be based on biopsies taken at 2 weeks.
The mean lamina propria mucosa (LPM) response in stool at week 2 will be compared between the two groups with Student's t test. | 2 weeks
  This will be based on biopsies taken at 2 weeks.
The mean C-reactive protein (CRP) at week 2 will be compared between the two groups with Student's t test. | 2 weeks
  Blood test checked at 2 weeks
The mean Fecal Calprotectin (FCP) at week 2 will be compared between the two groups with Student's t test. | 2 weeks
  Stool test checked at week 2
The mean lactulose to mannitol ratio (L/M) at week 2 will be compared between the two groups with Student's t test. | 2 weeks
  Urine test checked at week 2
The mean CRP at week 25 will be compared between the two groups with Student's t test. | 25 weeks
  Blood test checked at week 25
The mean FCP at week 25 will be compared between the two groups with Student's t test. | 25 weeks
  Stool test checked at week 25
The mean L/M ratio at week 25 will be compared between the two groups with Student's t test. | 25 weeks
  Urine test checked at week 25
The mean Crohn's Disease Activity Index (CDAI) scores calculated by study team at week 25 will be compared between the two groups with Student's t test | 2 weeks
  This score is based on blood tests, weight, and extra intestinal manifestations. The higher the score the worse the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Higgins, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No